CLINICAL TRIAL: NCT04461275
Title: ERAS 2.0 - Accelerated 23-hour ERAS Care for Colorectal Surgery
Brief Title: CHASE : aCcelerated 23-Hour erAS Care for Colorectal Surgery
Acronym: CHASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Z20202017
Record Dates: First submitted 2020-06-25; First posted 2020-07-08 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer; Enhanced Recovery After Surgery
Keywords: Colorectal Cancer; Enhanced Recovery After Surgery; Accelerated Care; Truly Minimally Invasive Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is an investigator-initiated, single-center prospective feasibility study. This feasibility study will compare 30 consecutive patients following the ERAS 2.0 program to 30 patients of a retrospective cohort who followed the current standard ERAS 1.0 protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERAS 2.0 group (Experimental): Patients included in the ERAS 2.0 group will follow the ERAS 2.0 accelerated care protocol.
  Interventions: Other: ERAS 2.0

INTERVENTIONS:
Other: ERAS 2.0 — ERAS 2.0 accelerated protocol with adequate fluid management, pain control and truly minimally invasive surgery (intracorporeal anastomosis)

SUMMARY:
Rationale: Throughout the years, there has been a rapid change in the perioperative protocols and procedures surrounding colorectal surgery. Upon the introduction of the Enhanced Recovery After Surgery (ERAS) program in Western countries, an improvement in postoperative outcomes was seen. Nowadays, researchers focus on further improving the current standard ERAS programs enabling an accelerated version hereof.

Objective: The aim of this study is to investigate the feasibility and safety of a 23-hour accelerated ERAS protocol (ERAS 2.0) for patients undergoing colorectal surgery compared to a retrospective cohort of patients who followed ERAS 1.0 for colorectal surgery. In this ERAS 2.0 protocol, patients undergoing colorectal surgery will be discharged within 23 hours after surgery.

Study design: This study is an investigator-initiated, single-center prospective study.

Study population: Patients aged ≥ 18 years ≤ 80 undergoing surgical resection for colorectal pathology that meet the eligibility criteria will be invited to participate in this study.

Intervention: Adhering to a strict multidisciplinary and multifaceted ERAS 2.0 protocol, patients receiving elective colorectal surgery will be discharged 23-hours after surgery.

Main study parameters/endpoints: Rate of the successful and safe application of the 23-hour accelerated ERAS 2.0 protocol for patients undergoing elective colorectal surgery. Success rate will be measured in readmission rate and safety will be measured with rate of serious adverse events (Clavien Dindo ≥3b). Success rate (feasibility) will also be measured in percentage of patients who were not able to be discharged 23 hours after surgery.

DETAILED DESCRIPTION:
The aim of this study is to investigate the feasibility and safety of a 23-hour accelerated ERAS 2.0 protocol for patients undergoing colorectal surgery compared to a retrospective cohort of patients who followed ERAS 1.0 for colorectal surgery. In this ERAS 2.0 protocol, patients undergoing colorectal surgery will be discharged within 23 hours after surgery.

Primary Objective:

To assess the successful and safe application of the 23-hour accelerated ERAS 2.0 protocol for patients undergoing colorectal surgery.

Secondary Objective(s):

* Postoperative outcomes, including morbidity and mortality within 30 days;
* Patient experience and satisfaction.

This study is an investigator-initiated, single-center prospective feasibility study. This feasibility study will compare 30 consecutive patients following the ERAS 2.0 program to 30 patients of a retrospective cohort who followed the current standard ERAS 1.0 protocol in Zuyderland Medical Center.

Population:

Patients diagnosed with malignant colorectal disease which requires surgical resection that meets the eligibility criteria will be invited to participate in this feasibility study. Patients will be approached on the surgical outpatient clinic at both locations from Zuyderland Medical Center. The study and actual surgery will take place only at location Sittard-Geleen.

Screening:

After written informed consent is obtained, participants are screened for further suitability. All participants will undergo a brief physical screening performed by an anesthesiologist. This screening will include: a complete cardiopulmonary physical examination, rest-EKG and routine laboratory workup. Should any contraindications be found during this screening, this will be used to further exclude patients from this study. In addition, participants are given extra information about ERAS 2.0 and expectations will be managed by discussing common side-effects and symptoms after general anesthesia and laparoscopic colorectal surgery.Only participants scheduled to undergo left-sided colorectal surgery are given a prescription for Bisacodyl 5mg as bowel preparation. Patients will be instructed to take 2 tablets the night before surgery and one tablet the morning of the surgery. Non-diabetic participants will be provided with 2 preoperative carbohydrate drinks (PreOp).

6.2.2 Preoperative Surgical ward On the day of surgery, participants are admitted early on the surgical ward and are prepared for surgery. They are required to present themselves at the surgical ward two hours prior to surgery. Participants will then be instructed to take the second preoperative carbohydrate drink (PreOp). Diabetic participants will not be provided with PreOp. As part of ERAS 2.0, it will be required of the participants to walk to the Holding with their bed with the assistance of their nurse.

Pre Anesthesia Care Unit (PACU) While participants are being prepared for anesthesia and surgery, they will once more be informed about the possible side-effects and discomfort associated with anesthesia and abdominal surgery. This in an effort to further manage expectations.

Preoperative administration of multimodal analgesia regimen is initiated in the PACU. This will consist of 1 gram Paracetamol and 600 milligrams Gabapentin (300 mg if GFR <60 ml/min or age> 70 years) intravenously.

Perioperative Participants are brought to the operating theater and the "time-out" check will be done. Here after the participant is prepared for anesthesia and surgery. Standard monitoring according to ASA guidelines will be applied.

Anesthesia Pre-induction: Spinal anesthesia consisting of 12.5 mg Bupivacaine combined with intrathecal morphine 300 mcg will be administered intravenously.

Induction: 1-2 mg per kg Propofol 2% plus TIVA (a mix of 50ml propofol plus 2% 500mcg Ultiva) at 4mcg/ml. In addition a bolus of Ketanest-S will be administered at 0.25 mg/kg. Dosages are adjusted to age and weight of the participant.

Fluid therapy: only balanced crystalloids are chosen for intravenous fluids (Ringer Lactate or Stereofundin). Optimization of fluid therapy is achieved by guided Esophageal Doppler or Flo Trac System management up until the end of surgery. Continuous perfusion of Ringer Lactate / Stereofundin will be set at 3 ml/kg/hour IV.

Ventilation: Optimal ventilation parameters will be obtained during surgery with: Total Volume 6-8 ml/kg; minimum FiO2 to prevent atelectasis and optimal PEEP (patients specific) to prevent peri- and postoperative atelectasis.

Surgery - peroperative All participants will be operated on laparoscopically, in a true minimally invasive manner. With exception of the following two factors pertaining to ERAS 2.0, all operations will be performed according to standard hospital protocols. (1) Starting intra-abdominal pressure will be set at 12 mmHg. During surgery, the intra-abdominal pressure will be gradually reduced to an end pressure of 8 mmHg. This method has been proven to be safe and is associated with less postoperative pain caused by laparoscopic insufflation. (2) Primary anastomosis will be performed intracorporeally as this method is associated with similar results to extracorporeal anastomosis. No additional mini-laparotomy will be performed. The specimen will be extracted through a suprapubic pfannenstiel incision. After surgery, routine postoperative measures will be used to omit sedation and commence recovery. If surgery was uncomplicated and performed under 2 hours, the urinary catheter will be removed in the operation theater.

Postoperative Recovery ward After surgery, participants are brought to the recovery ward where further care will be given before transporting them to the surgical ward. Here participants are continuously monitored and checked for postoperative nausea, pain and discomfort. In case of nausea and/or vomiting, participants are treated according to standard hospital protocols. To bridge postoperative pain management, participants will receive 7.5mg Meloxicam postoperatively. Postoperative pain management consists of 1000mg Paracetamol IV every 6 hours. If necessary, 5-20mg Oxynorm (tablet) can be offered up to 6 times a day. To stimulate intake and gastrointestinal motility, patients are offered a popsicle on the recovery ward.

Surgical ward

Postoperative day 0:

Upon arrival on the surgical ward, postoperative care is resumed according to standard hospital protocol with respect to anti-emetic care, patient monitoring and thromboprophylaxis. Routine physical examination and evaluation will take place.

The postoperative care-points of ERAS 2.0 are: Minimal-opiate pain management; early removal of the urinary catheter, early oral intake; early stop of IV-fluids and early mobilization. Pain management is achieved with Paracetamol and Meloxicam, and if needed Oxynorm. Standard hospital dosages will be used. At 22:00 hours, if still in situ, urinary catheters will be removed. Intake is stimulated and participants will be offered food and beverages, starting with fluids gradually increasing to full oral intake tolerance of their normal diet. Participants are encouraged to sit up straight in bed as much as possible and to mobilize in their room.

Postoperative day 1:

The following day, participants will be evaluated for measure of recovery and suitability for discharge. Routine physical examination and evaluation will take place. The surgical incision sites will be evaluated and the abdomen will be examined for swelling, redness and for possible hematoma/bleeds. Participants will be evaluated for pain using the VAS pain score and will be evaluated for other signs of discomfort.

Participants are considered as ' functionally recovered' and safe for discharge if the following criteria are met:

* Pain under control with oral analgesics (VAS <4)
* No symptoms of nausea and/or vomiting
* Flatus or passing of stools
* Oral intake possible (resumed full diet)
* Spontaneous micturition
* Able to mobilize independently
* No alarm signs present (fever, tachycardia, hypotension, dyspnea or somnolence).

Participants are only discharged if they tick off all the requirements on the discharge checklist. Before discharge, their nurse will explain the recovery trajectory after discharge, including the telephonic aftercare. This includes pain management, dietary and mobilizing advice, thromboprophylaxis instructions and alarm symptoms to be weary of. Participants will receive a discharge folder with all necessary information, including all available contact numbers. The abovementioned information will be included in the discharge letter that patients receive upon leaving the surgical ward.

Care after discharge Telephonic aftercare On the evening of the day of discharge, participants will be contacted by the attending nurse. A premade ERAS 2.0 checklist concerning recovery and possible alarm symptoms will be used to assess recovery. On postoperative day 4, participants will be contacted again via telephone by the attending nurse practitioner, and the same steps are repeated.

Outpatient clinic Participants are given an appointment with a colorectal surgeon to be checked at the surgical outpatient clinic. During this appointment, the overall experience of the participant will be evaluated, together with his/her clinical recovery. The participant will be provided with an evaluation form.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Is ≥ 18 years ≤ 80;
* BMI ≤ 35 kg/m2;
* WHO performance status = 0
* Is diagnosed with (non-complicated) colorectal cancer
* Is scheduled to undergo elective laparoscopic colorectal surgery (ileocecal resection, right or left hemicolectomy, transvers colon resection) with primary anastomosis;
* Primary anastomosis is performed intracorporeally;
* Uncomplicated operation;
* Readily available ambulant care provided by an adult family member for the first 24 hours after discharge;
* Patient is adequately reachable by phone.

Exclusion Criteria:

* ASA classification ≥ 3;
* Subjects who have limited mobility and/or need to be aided/assisted when mobilizing;
* Subjects with a history of active pulmonary infection, any other active infection, any uncontrolled medical disease
* Subjects with a contraindication for oral NSAIDs;
* Subjects with a contraindication for spinal anesthesia;
* Subjects requiring parenteral nutrition prior to surgery;
* Subjects scheduled to undergo lower rectal resections;
* Subjects receiving an ostomy;
* Subjects who experience complications preoperatively;
* Subjects who are mentally incompetent, challenged or requiring aid with daily life activities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of the successful and safe application of the 23-hour accelerated ERAS 2.0 protocol for patients undergoing elective colorectal surgery. | 30 days
  Success rate (feasibility) will be measured in readmission rate and safety will be measured with rate of serious adverse events (Clavien Dindo ≥3b).

SECONDARY OUTCOMES:
• Number of Participants who develop Postoperative Complications within 30 days | 30 day
  • Number of Participants who develop Postoperative Complications within 30 days
• Number of Participants with Postoperative Mortality within 30 days | 30 days
  • Number of Participants with Postoperative Mortality within 30 days
• Patient satisfaction evaluation by means of a questionnaire to evaluate the patients subjective experience during the duration of this study. | 10 days
  • Patient satisfaction evaluation questionnaire to evaluate the patients subjective experience during the duration of this study and their subjective experience with the ERAS 2.0 protocol. In this questionnaire, patients will be asked to evaluate their experience based on 5 pre-set questions with a 10-point scale (1 being very bad and 10 being very good).
  1. Were you sufficiently informed about the ERAS 2.0 protocol?
  2. How did you experience the guidance provided (by nurses and doctors) within this protocol?
  3. Was the care provided after hospital discharge satisfactory?
  4. Was it necessary to contact the hospital after discharge? And if yes, how often?
  5. What grade would you give this programme?

OTHER OUTCOMES:
• Demographic parameters | Upon inclusion
  • Demographic parameters such as age, height, sex, comorbidities
• Disease related demographics | After surgery and within 14 days after surgery
  • Disease related demographics such as tumor type, location, type of resection, etc.
• Short Nutritional Assessment Questionnaire (SNAQ) | Upon inclusion
  • Short Nutritional Assessment Questionnaire (SNAQ) Lowest score: 0 and Highest score: 5
  score 0 or 1: low risk of malnutrition score 2: moderate risk of malnutrition score ≥ 3: high risk of malnutrition, refer to dietician
• Groningen Frailty Index (GFI) | Upon inclusion
  • Groningen Frailty Index (GFI)
  Lowest score: 0 and Highest score: 15
  score <4: not frail score 4-5: frail score ≥ 6: really frail

CONTACTS AND LOCATIONS:
Overall Officials: James van Bastelaar, M.D., PhD, Principal Investigator — GE-, Oncologic-surgeon
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Mazrou AM, Chiuzan C, Kiran RP. Factors influencing discharge disposition after colectomy. Surg Endosc. 2018 Jul;32(7):3032-3040. doi: 10.1007/s00464-017-6013-z. Epub 2017 Dec 27. PMID 29282575
- [Background] Dobradin A, Ganji M, Alam SE, Kar PM. Laparoscopic colon resections with discharge less than 24 hours. JSLS. 2013 Apr-Jun;17(2):198-203. doi: 10.4293/108680813X13654754535791. PMID 23925012
- [Background] Chand M, De'Ath HD, Rasheed S, Mehta C, Bromilow J, Qureshi T. The influence of peri-operative factors for accelerated discharge following laparoscopic colorectal surgery when combined with an enhanced recovery after surgery (ERAS) pathway. Int J Surg. 2016 Jan;25:59-63. doi: 10.1016/j.ijsu.2015.11.047. Epub 2015 Nov 30. PMID 26654893
- [Result] Rossi G, Vaccarezza H, Vaccaro CA, Mentz RE, Im V, Alvarez A, Quintana GO. Two-day hospital stay after laparoscopic colorectal surgery under an enhanced recovery after surgery (ERAS) pathway. World J Surg. 2013 Oct;37(10):2483-9. doi: 10.1007/s00268-013-2155-x. PMID 23881088
- [Result] Emmanuel A, Chohda E, Botfield C, Ellul J. Accelerated discharge within 72 hours of colorectal cancer resection using simple discharge criteria. Ann R Coll Surg Engl. 2018 Jan;100(1):52-56. doi: 10.1308/rcsann.2017.0149. Epub 2017 Sep 15. PMID 29022790
- [Result] Levy BF, Scott MJ, Fawcett WJ, Rockall TA. 23-hour-stay laparoscopic colectomy. Dis Colon Rectum. 2009 Jul;52(7):1239-43. doi: 10.1007/DCR.0b013e3181a0b32d. PMID 19571699